CLINICAL TRIAL: NCT05745974
Title: Post COVID-19 Complications in Children Attending Assiut University Children Hospital
Brief Title: Post COVID-19 Complications in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Gamal Ali, physician, Assiut University
Other Study IDs: Post COVID-19 complications
Record Dates: First submitted 2023-02-23; First posted 2023-02-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Post COVID-19 Condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lymphocytic count — taking blood samples and COVID-19 swab
  Other Names: C-Reactive Protein; serum ferritin; D dimer; RT PCR for COVID-19

SUMMARY:
Is to record post COVID-19 complications in patients below 18 years old in assiut University children hospital

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is one of the largest public health pandemics since the Spanish flu of1918. With a wide spectrum of clinical manifestations, COVID-19 has caused major setbacks in healthcare worldwide and challenged the capabilities of some of the most accomplished health care systems in the world. Although up to 80% of patients are initially asymptomatic, a nonnegligible percentage eventually require hospitalization and intensive care admission (ICU)Johns Hopkins,2020.Currently, the worst complication of COVID-19 is vascular inflammation and degeneration, AbdelMassih AF, Kamel A et al. Most children with COVID-19 present with a range of signs and symptoms that are not severe or specific enough to prompt disease testing.3 Some children and adolescents show no symptoms at all,Han MS, Choi EH, et al .The challenge with unrecognized COVID-19 cases is that asymptomatic children might become silent carriers in the community, DeBiasi RL, Delaney M,et al.or be at risk of developing post-COVID-19 complications. post-acute COVID-19 includes patients with persistent or delayed symptoms that develop, or last, more than 3 weeks after symptom-onset. The 3-week period is in line with evidence that viable virus is rarely detected past 10 days in mild to moderate COVID-19, and rarely past 20 days in severe cases, DeBiasi RL, Delaney M, et al. Another term used to describe this condition is "long COVID". Butler M, Pollak TA, Baker HA,et al. Since MIS-C is not true sequelae, we will report on MIS-C separately from post-acute COVID-19. MIS-C is a newl recognized illness associated with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. McMurray et al. (2020) described MIS-C as a post-viral systemic inflammatory vasculopathy of children following SARS-CoV-2 infection, with similar clinical presentations to Kawasaki disease. Ontario Agency for Health Protection and Promotion,2020. In April 2020, reports from the United Kingdom documented a clinical presentation in children identical to Kawasaki disease (KD) or toxic shock syndrome. Since then, there has been an increase in reported cases of similarly affected children in other parts of the wothe, Riphagen S, Gomez X, et al ,2020. The cases have been reported from Asia, North America, Latin America and Europe in the past 3 months, describing children with COVID-19-associated multisystem inflammatory syndrome in children (MIS-C), which is likely to develop after the disease instead of developing during the acute phase of COVID-19 Jones VG, Mills M, et al, 2020.Thrombotic complications have alsobeen reported in children with COVID-19, Mitchell W, Davilla J, Whitworth H, Sartain SE,2020.

ELIGIBILITY:
Inclusion Criteria:

* Patients below 18 years of age
* Patients who are Tested swab positive for COVID-19
* New cases that will be tested swab positive for COVID-19
* Pateints who are suspected of kawazaki disease

Exclusion Criteria:

* Patients above 18 years
* Patients having psychological disorders patients having chronic disease like cardiac, chest , and renal diseases

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children below 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-24 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
record post COVID-19 complications in patients below 18 years old | Baseline
  detection of any complications related to post infection with COVID-19 by using the laboratory investigations

REFERENCES:
- [Background] Whitworth H, Sartain SE, Kumar R, Armstrong K, Ballester L, Betensky M, Cohen CT, Diaz R, Diorio C, Goldenberg NA, Jaffray J, Keegan J, Malone K, Randolph AG, Rifkin-Zenenberg S, Leung WS, Sochet A, Srivaths L, Zia A, Raffini L. Rate of thrombosis in children and adolescents hospitalized with COVID-19 or MIS-C. Blood. 2021 Jul 15;138(2):190-198. doi: 10.1182/blood.2020010218. PMID 33895804
- [Result] AbdelMassih AF, Kamel A, Mishriky F, Ismail HA, El Qadi L, Malak L, El-Husseiny M, Ashraf M, Hafez N, AlShehry N, El-Husseiny N, AbdelRaouf N, Shebl N, Hafez N, Youssef N, Afdal P, Hozaien R, Menshawey R, Saeed R, Fouda R. Is it infection or rather vascular inflammation? Game-changer insights and recommendations from patterns of multi-organ involvement and affected subgroups in COVID-19. Cardiovasc Endocrinol Metab. 2020 Jun 11;9(3):110-120. doi: 10.1097/XCE.0000000000000211. eCollection 2020 Sep. PMID 32803145
- [Result] Han MS, Choi EH, Chang SH, Jin BL, Lee EJ, Kim BN, Kim MK, Doo K, Seo JH, Kim YJ, Kim YJ, Park JY, Suh SB, Lee H, Cho EY, Kim DH, Kim JM, Kim HY, Park SE, Lee JK, Jo DS, Cho SM, Choi JH, Jo KJ, Choe YJ, Kim KH, Kim JH. Clinical Characteristics and Viral RNA Detection in Children With Coronavirus Disease 2019 in the Republic of Korea. JAMA Pediatr. 2021 Jan 1;175(1):73-80. doi: 10.1001/jamapediatrics.2020.3988. PMID 32857112
- [Result] DeBiasi RL, Delaney M. Symptomatic and Asymptomatic Viral Shedding in Pediatric Patients Infected With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2): Under the Surface. JAMA Pediatr. 2021 Jan 1;175(1):16-18. doi: 10.1001/jamapediatrics.2020.3996. No abstract available. PMID 32857158
- [Result] Butler M, Pollak TA, Rooney AG, Michael BD, Nicholson TR. Neuropsychiatric complications of covid-19. BMJ. 2020 Oct 13;371:m3871. doi: 10.1136/bmj.m3871. No abstract available. PMID 33051183
- [Result] Baker HA, Safavynia SA, Evered LA. The 'third wave': impending cognitive and functional decline in COVID-19 survivors. Br J Anaesth. 2021 Jan;126(1):44-47. doi: 10.1016/j.bja.2020.09.045. Epub 2020 Oct 21. No abstract available. PMID 33187638
- [Result] McMurray JC, May JW, Cunningham MW, Jones OY. Multisystem Inflammatory Syndrome in Children (MIS-C), a Post-viral Myocarditis and Systemic Vasculitis-A Critical Review of Its Pathogenesis and Treatment. Front Pediatr. 2020 Dec 16;8:626182. doi: 10.3389/fped.2020.626182. eCollection 2020. PMID 33425823
- [Result] Riphagen S, Gomez X, Gonzalez-Martinez C, Wilkinson N, Theocharis P. Hyperinflammatory shock in children during COVID-19 pandemic. Lancet. 2020 May 23;395(10237):1607-1608. doi: 10.1016/S0140-6736(20)31094-1. Epub 2020 May 7. No abstract available. PMID 32386565
- [Result] Jones VG, Mills M, Suarez D, Hogan CA, Yeh D, Segal JB, Nguyen EL, Barsh GR, Maskatia S, Mathew R. COVID-19 and Kawasaki Disease: Novel Virus and Novel Case. Hosp Pediatr. 2020 Jun;10(6):537-540. doi: 10.1542/hpeds.2020-0123. Epub 2020 Apr 7. PMID 32265235
- [Result] Mitchell WB, Davila J, Keenan J, Jackson J, Tal A, Morrone KA, Silver EJ, O'Brien S, Manwani D. Children and young adults hospitalized for severe COVID-19 exhibit thrombotic coagulopathy. Pediatr Blood Cancer. 2021 Jul;68(7):e28975. doi: 10.1002/pbc.28975. Epub 2021 Mar 4. PMID 33661561